CLINICAL TRIAL: NCT06245187
Title: Get With the Guidelines-Atrial Fibrillation
Brief Title: Get With the Guidelines Atrial Fibrillation Registry
Acronym: GWTG-AF
Status: Recruiting | Type: Observational
Sponsor: American Heart Association (Other)
Responsible Party: Sponsor
Other Study IDs: 002
Record Dates: First submitted 2016-02-23; First posted 2024-02-07 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-01

CONDITIONS: Atrial Fibrillation; Atrial Flutter
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: GWTG Atrial Fibrillation program — Evidence based recommended therapies and counseling prior to hospital discharge.

SUMMARY:
Get With The Guidelines-Atrial Fibrillation is designed to assist hospital care teams in consistently providing the latest evidence-based treatment for their AFib patients. At the same time, it offers a means of monitoring the quality of AFib care in U.S. hospitals and building a database for continued research and further quality improvement.

DETAILED DESCRIPTION:
Get With The Guidelines-Atrial Fibrillation was initiated in 2013 with over 88 U.S. hospitals participating is designed to assist hospital care teams in consistently providing the latest evidence-based treatment for their AFib patients. At the same time, it offers a means of monitoring the quality of AFib care in U.S. hospitals and building a database for continued research and further quality improvement.

Achievement measures tracked through Get With The Guidelines-Atrial Fibrillation:

1. ACEI/ARB at discharge for LVSD
2. Assessment of thromboembolic risk factors
3. Beta Blocker at discharge
4. Discharged on FDA-approved anticoagulation therapy
5. PT/INR planned follow-up
6. Statin at discharge in AF patients with CAD, CVA/TIA or PVD.

Quality measures tracked through Get With The Guidelines-Atrial Fibrillation:

1. Aldosterone antagonist at discharge
2. Atrial fibrillation patient education
3. Anticoagulation therapy education
4. CHA2DS2-VASC reported
5. Discharge heart rate <110bpm
6. Smoking cessation
7. Warfarin at discharge for valvular atrial fibrillation

Additional measures collected by Get With The Guidelines-Atrial Fibrillation can be viewed at: http://www.heart.org/idc/groups/heart-public/@private/@wcm/@hcm/@gwtg/documents/downloadable/ucm_451183.pdf

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized with nonvalvular Atrial Fibrillation or Atrial Flutter

Exclusion Criteria:

* Patients who do not have nonvalvular Atrial Fibrillation or Atrial Flutter
* Patients under 18 years of age
* Patients not admitted as inpatients.
* Patients on comfort care only
* Patients discharged to hospice.

Ages: 18 Years to 125 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is patients with the diagnosis of nonvalvular Atrial Fibrillation or Atrial Flutter.
Sampling Method: Probability Sample
Enrollment: 17198 (Estimated)
Dates: Start 2013-01; Primary Completion 2040-01 (Estimated); Study Completion 2040-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac Tamponade and/or Pericardiocentesis Following Ablation | 30 days
  Percent of patients with cardiac tamponade and/or pericardiocentesis occurring within 30 days following ablation procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Javed Butler, MD, Principal Investigator — American Heart Association
Locations (1):
- Amy Bennett, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC Jr, Conti JB, Ellinor PT, Ezekowitz MD, Field ME, Murray KT, Sacco RL, Stevenson WG, Tchou PJ, Tracy CM, Yancy CW; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2014 Dec 2;64(21):e1-76. doi: 10.1016/j.jacc.2014.03.022. Epub 2014 Mar 28. No abstract available. PMID 24685669